CLINICAL TRIAL: NCT00862160
Title: Acute Cerebrovascular Events During Extracorporeal Circulation a Comparison of New Minimized Perfusion Circuit to Standard Cardiopulmonary Bypass
Brief Title: Incidence of Acute Cerebrovascular Events Using Either Minimized or Standard Cardiopulmonary Bypass Circuit
Acronym: ROCsafeTM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Academic Teaching Hospital Braunschweig (Other); Terumo Europe N.V. (Industry)
Responsible Party: PD Dr. med. Ingo Kutschka, HannoverMS, Clinic of Cardiac Thoracic Transplantation and Vascular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T201E1
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Coronary Artery Disease; Acute Cerebrovascular Accident; Intracranial Embolism; Embolism, Air
Keywords: coronary artery bypass surgery; cardiopulmonary bypass; heart lung machine; acute cerebrovascular event; intracranial embolism; embolism, air; outcome assessment (health care); neuropsychological tests; magnetic resonance imaging; saccadic eye movement test
MeSH Terms: conditions — Coronary Artery Disease; Stroke; Intracranial Embolism; Embolism, Air

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): using minimized cardiopulmonary bypass circuit ROCsafeTM
  Interventions: Device: ROCsafeTM
- 2 (No Intervention): using standard cardiopulmonary bypass circuit

INTERVENTIONS:
Device: ROCsafeTM — using minimized perfusion circuit while CABG
  Arms: 1

SUMMARY:
The prospective, randomized, two centre study investigates acute cerebrovascular events during extracorporal circulation and the early post operative outcome when using either the minimized cardiopulmonary bypass circuit (ROCsafeTM) or a standard cardiopulmonary bypass circuit in patients undergoing coronary artery bypass grafting.

DETAILED DESCRIPTION:
Coronary artery bypass grafting with extracorporal circulation is established as the golden standard. The conventional cardiopulmonary bypass (CPB) system is associated with inflammatory reaction, hemolysis, hemodilution an disturbances of the blood coagulation system. Also it's well known that neurological disturbances caused by embolic material and air bubbles are potential risks of CPB. The new minimized perfusion circuit ROCsafeTM is a closed, reservoir-less, reduced prime, surface coated circuit, with optimized safety features in effectively eliminate both macro and micro air bubbles and should optimize the clinical outcome after CABG using cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 17 years
* Patient is acceptable candidate for CABG operation
* Patient or the patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* Ejection fraction less than 30 %
* Valve surgery
* Acute endocarditis or history of endocarditis
* Cerebral ischemia within 4 weeks before surgery
* Detection of intracardial thrombi in preoperative echocardiography
* Stenosis of A. carotis int. greater than 70 %
* Patients older than 80 years
* Patients on dialysis
* Acute myocardial ischemia or infarction within two weeks before inclusion
* Markedly elevated baseline C-reactive protein (CRP) or leucocytosis
* Cancer or immunologic diseases
* Dysregulation of the coagulation cascade (not concerning INR or PTT under cumarin or heparin treatment)
* Intake of steroids or NSAR
* Female of childbearing potential
* Participation in an other study
* Contraindication for MRI (e.g. pacemaker, any kind of implanted metal)
* Claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
fresh micro-lesions in cranial MRT | before and 72 h after CABG

SECONDARY OUTCOMES:
Death | 30 days after CABG
Neurological events | between CABG and discharge
Neurocognitive function | before and 3-4 days after CABG and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Kutschka, PD Dr. med., Principal Investigator — Hannover Medical School
Locations (2):
- Germany (2):
  - Klinikum Braunschweig, Department of Cardiothoracic Surgery, Braunschweig
  - Hannover Medical School, Clinic for Cardiac, Thoracic, Transplantation and Vascular Surgery, Hanover